CLINICAL TRIAL: NCT05678478
Title: Perceptions,Social Representations and Experience of Lyme Borreliosis and Ticks in Adolescents Likely to be Infected and Their Parents
Acronym: ADO-LY
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: ADO-LY
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Lyme Disease
MeSH Terms: conditions — Lyme Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: semi-directed interview concerning the experience of adolescents and their parents on Lyme borreliosis and on the tick. — semi-structured interview on the experience of adolescents and their parents on Lyme borreliosis and the tick.
  The interviews will be semi-directed in physical presence. Three interviews will be conducted.
  The minor will be questioned first, then the parent(s). And finally, the whole family in one interview. All interviews will be audio recorded with parallel note taking in order to best transcribe the visual expressions. The interviews will be transcribed in writing and pseudonymised.

SUMMARY:
the study is offered to adolescents aged 12 to 17 and their families suspected of or suffering from Lyme barilliosis.

During inclusion, three interviews will be carried out for each family. This choice of the number of interviews per family seems the most appropriate to have a plurality of answers to the questions asked. Thus, these will have a duration of 30 min to 1 hour and will be carried out by an anthropologist. The first interview will be with the teenager. The second interview will then concern the parent(s). Finally, the last appointment will be with the teenager and his parents.

DETAILED DESCRIPTION:
the study is offered to adolescents aged 12 to 17 and their families suspected of or suffering from Lyme barilliosis.

During inclusion, three interviews will be carried out for each family. This choice of the number of interviews per family seems the most appropriate to have a plurality of answers to the questions asked. Thus, these will have a duration of 30 min to 1 hour and will be carried out by an anthropologist. The first interview will be with the teenager. The second interview will then concern the parent(s). Finally, the last appointment will be with the teenager and his parents.

After a few introductory questions concerning the socio-demographic characteristics of adolescents, their medical history and their exposure to ticks, the anthropologist will ask the semi-open questions.

As for the parent(s), the anthropologist will ask them questions directly related to Lyme borreliosis and the tick. Finally, questions will be proposed simultaneously during a joint interview with the teenager and his parents.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 12 years old and maximum 17 years old.
* Be accompanied by a holder of parental authority
* Live in metropolitan France.
* Suspect or have Lyme borreliosis
* Non-objection for participation in the protocol

Exclusion Criteria:

* Refusal of participation of a holder of parental authority and of the adolescent
* Non-mastery of oral French by the teenager or his parents
* Protected persons (patients under guardianship or curatorship, pregnant or nursing women, persons deprived of liberty, person unable to express their non-objection)

Ages: 12 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: These are patients aged 12 to 17 years maximum and their parents come for a suspicion of adolescent Lyme borreliosis.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Story of the teenager and one of his parents or both parents | Baseline
  analysis and identification of perceptions, representations and experiences of adolescents and their parents on Lyme borreliosis and ticks

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Intercommunal Villeneuve Saint Georges, Crosne
  - Hôpital Armand Trousseau AP-HP, Paris

IPD SHARING:
Plan to Share IPD: No